CLINICAL TRIAL: NCT07217249
Title: Diabetes Endothelial Keratoplasty Study (DEKS): Impact of Diabetes and Other Predictors on Corneal Transplant Endothelial Cell Loss and Success
Brief Title: Effect of Donor Diabetes and Other Factors on Corneal Transplant Endothelial Cell Loss and Success at 5 Years
Acronym: DEKS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEKS 5-year Extension Study; 1UG1EY037206-01 (NIH); 5UG1EY030030-05 (NIH)
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Fuchs Endothelial Corneal Dystrophy; Corneal Endothelial Decompensation
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned cornea from a donor without diabetes (Active Comparator): Eyes assigned to this arm receive a cornea from a donor without diabetes and undergo Descemet membrane endothelial keratoplasty.
  Interventions: Procedure: Descemet membrane endothelial keratoplasty
- Assigned cornea from a donor with diabetes (Active Comparator): Eyes assigned to this arm receive a cornea from a donor with diabetes for Descemet membrane endothelial keratoplasty.
  Interventions: Procedure: Descemet membrane endothelial keratoplasty

INTERVENTIONS:
Procedure: Descemet membrane endothelial keratoplasty — Replacement of the recipient corneal endothelial and Descemet membrane with healthy tissue from a donor cornea.

SUMMARY:
This multi-center clinical trial is designed to assess the association of diabetes in a cornea donor with transplant success and loss of endothelial cells 5 years following Descemet membrane endothelial keratoplasty (DMEK). Study eyes are assigned to receive either a cornea from a donor without diabetes or a cornea from a donor with diabetes in a masked fashion.

ELIGIBILITY:
Inclusion Criteria:

* Willing to return to the study site for follow up at 3 and 5 years after a Descemet membrane endothelial keratoplasty procedure
* Fluent in English or Spanish
* Willing to have fingerstick blood sample collected to determine HbA1c level
* Participated and completed 12-month follow-up in the DEKS study for one or both eyes or a DEKS participant that had a study eye regraft prior to the 12-month visit.

Exclusion Criteria:

* Lack cognitive capacity such that consent could not be provided.

Ages: 30 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2029-12-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in central corneal endothelial cell density 5 years after Descemet membrane endothelial keratoplasty. | Subjects are followed for 5 years after corneal transplantation.
  Central corneal endothelial cell density will be assessed by specular microscopy at 3 and 5 years after Descemet membrane endothelial keratoplasty and the results will be compared with the baseline donor endothelial cell density assessed at the eye bank that provided the donor tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lass, MD, Principal Investigator — Case Western Reserve University
Locations (14):
- United States (14):
  - Georgia Eye Partners, Atlanta, Georgia
  - Price Vision Group, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Kansas City Eye Clinic, Overland Park, Kansas
  - Huffman and Huffman, PSC, Lexington, Kentucky
  - Mid-Atlantic Cornea Consultants, Baltimore, Maryland
  - The Wilmer Eye Institute/Johns Hopkins, Baltimore, Maryland
  - University of Michigan/Kellogg Eye Center, Ann Arbor, Michigan
  - Verdier Eye Center, Grand Rapids, Michigan
  - Minnesota Eye Consultants, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Associated Eye Care, Stillwater, Minnesota
  - Moyes Eye Center, Kansas City, Missouri
  - Legacy Devers Eye Institute, Portland, Oregon